#### NCT04206293

Study ID: CMO-MA-FAS-0617

**Title:** Prospective, Open-Label Study, to Evaluate The Impact on Skin Quality Attributes by Juvederm® Volite Injection on Healthy Volunteers

Statistical Analysis Plan Date: 16Jan2020

# STATISTICAL ANALYSIS PLAN



# PROSPECTIVE, OPEN-LABEL STUDY, TO EVALUATE THE IMPACT ON SKIN QUALITY ATTRIBUTES BY JUVEDERM® VOLITE INJECTION ON HEALTHY VOLUNTEERS

Protocol #: 18E2581

| Investigational product: | Juvederm® VOLITE |
|---|---|
| Forms: | Sterile gel |
| Administration | Intradermal injection |
| CRO | DERMSCAN - Pharmascan<br>114 Boulevard du 11 Novembre 1918<br>69100 VILLEURBANNE<br>FRANCE |
| Study centres Dermscan Poland Sp. z o.o. ul. Matuszewskiego 12 80-288 GDANSK POLAND | |
| Principal Investigators: | |
| Sponsor: | Allergan Pharmaceuticals International Limited Clonshaugh Industrial Estate Coolock Dublin 17 Ireland |
| Date and version: | Final Version 1.0<br>16/01/2020 |
| Author of the report | Biostatistician: |

# **TABLE OF CONTENTS**

| 1. ( | OBJECTIVES | 5 |
|---|---|---|
| 2. 9 | SYNOPSIS OF THE PROTOCOL | 5 |
| 3. ( | OVERALL STUDY CONSIDERATIONS | <u>c</u> |
| 3.1 | | |
| 3.2 | | |
| 3.3 | | |
| 3.4 | | |
| 3.5 | | |
| 3.6 | | |
| 3.7 | | |
| 3 | 3.7.1. Performance outcomes | 11 |
| | 3.7.1.1. Summary of performance assessments | 11 |
| | 3.7.2. Safety outcomes | |
| 3 | | |
| | 3.7.2.1. Injection Site Reactions | |
| | 3.7.2.2. Other adverse events | |
| 4. 9 | STATISTICAL METHODOLOGY | 14 |
| 4.1 | L. DESCRIPTIVE ANALYSIS | 1/ |
| 4.1 | | |
| 4.3 | | |
| 4.4 | • | |
| 4.5 | | |
| 4.6 | | |
| 4.7 | | |
| 4.8 | | |
| 4.9 | | |
| 4.1 | · | |
| 4.1 | 11. STATISTICAL SOFTWARE | 15 |
| 5. 9 | STATISTICAL ANALYSIS | 15 |
| 5.1 | L. DEFINITION OF ANALYSIS POPULATION | 15 |
| 5.2 | | |
| 5.3 | | |
| 5.4 | | _ |
| 5.5 | | |
| | 5.5.1. Skin quality measurements | 1 <i>6</i> |
| 5.6 | 5. SAFETY EVALUATION | 18 |
| 6. 9 | SIGNATURES | 19 |
| | APPENDICES : STRUCTURE OF TABLES | |
| 7.1 | | |
| 7.2 | 2. Statistical table for summarizing quantitative data | |
| - | • | |
| 7.3 | , | |
| 7.3<br>7.4 | | |
| 7.4 | +. MUVENJE EVENIJO JINI NEJOJO | |



Allergan

# **LIST OF ABBREVIATIONS AND TERMS**

| A.U | Arbitrary Unite |
|------|----------------------------------|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| CI | Confidence interval |
| D | Day |
| GU | Glossymeter Units |
| IP | Investigational product |
| ISR | Injection Site Reaction |
| max | Maximum value |
| min | Minimum value |
| miss | Number of missing data |
| mm | Millimeter |
| N | Number of valid data |
| NRS | Numerial Rating Scale |
| PT | Preferred Term |
| Q1 | First quartile |
| Q3 | Third quartile |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SE | Standard error of estimated mean |
| SEM | Standard error of the mean |
| SOC | System Organ Class |
| TDC | Tissue Dielectric Constant |



Allergan

| Allergen | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| Allergan | PIOLOCOI # 18E2381PL | Date:16/01/2020 |

#### 1. OBJECTIVES

This statistical analysis plan (SAP) provides a detailed description of the statistics that will be performed on the efficacy and safety parameters and other data of the clinical study "PROSPECTIVE, OPEN-LABEL STUDY, TO EVALUATE THE IMPACT ON SKIN QUALITY ATTRIBUTES BY JUVEDERM® VOLITE INJECTION ON HEALTHY VOLUNTEERS" with the reference 18E2581PL – CMO-MA-FAS-0617

## 2. SYNOPSIS OF THE PROTOCOL

| Clinical investigation plan #: | 18E2581PL – CMO-MA-FAS-0617 |
|---|---|
| Title of the Clinical Investigation: | PROSPECTIVE, OPEN-LABEL STUDY, TO EVALUATE THE IMPACT ON SKIN QUALITY ATTRIBUTES BY JUVEDERM® VOLITE INJECTION ON HEALTHY VOLUNTEERS |
| Allergan Pharmaceuticals International Limited Clonshaugh Industrial Estate Sponsor: Coolock Dublin 17 Ireland | |
| Objectives: | To evaluate the impact on skin quality attributes, including physical measurements following administration of Juvéderm® VOLITE in the volar forearms of healthy volunteers |
| Design: | Prospective, single-center, open study |
| Planned Sample Size: | 11 subjects included for at least 10 subjects analyzed |
| Number of centres: | One center |
| Number of centres: 1. Healthy subject 2. Sex: male and female 3. Age: between 30 and 50 years old at the time of the written consent 4. Subjects with Fitzpatrick skin type II or III. 5. Subject willing to receive Juvéderm* VOLITE in the forearms and agrees to com required procedures, including having 6 punch biopsies taken in the forearms and (HIV, B and C hepatitis analysis at screening). | |
| Exclusion criteria: | In terms of population: |

| eurofins Dermscan Pharmascan | PRM03-F-198_EN_V2<br>STATISTICAL ANALYSIS PLAN | Page 5/27 |
|---|---|---|

1. Pregnant or nursing woman or planning a pregnancy during the study.

- 4. Subject participating to another research on human beings or being in an exclusion period for a previous study.
- 5. Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
- 6. Subject having other resorbable filling product injections, a laser treatment, an ultrasound-based treatment, radiation treatment, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the studied zones within the past 12 months prior to study start.
- 7. Subject with subcutaneous retaining structure on the studied zones (meshing, threads, gold strand).
- 8. Subject having received injections of permanent or semi-permanent filling products in the studied zones.



Related to previous or ongoing treatment



| Allorgon | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| Allergan | Protocol # 18E2581PL | Date:16/01/2020 |

- 24. Subject under anti-coagulant treatment or treatment liable to interfere with the healing process or hemostasis, during the previous month and during the study.
- 25. Subject receiving or is planning to receive anti-inflammatory drugs (oral/injectable corticosteroids or NSAIDs, e.g., aspirin, ibuprofen), or other substances known to increase coagulation time (herbal supplements with garlic or ginkgo biloba, etc) for 10 days prior to study treatment and 3 days after.
- 26. Subject under immunosuppressive therapy.

Investigational device:

Name / code: Juvéderm® VOLITE

Galenic form: Sterile gel in disposable syringe

**Dosage:** On Day 0 (D0) the specialist injector will treat the study area with an appropriate volume based

on his/her clinical experience and according to Instructions for Use.

**Administration route:** Intra-dermal injection in forearms

#### **Performance exploratory Endpoints**

Changes in skin quality parameters, one and three months after Juvéderm® VOLITE injection in the forearms, in comparison with before treatment (D0). Evaluated skin parameters and instruments used are summarized in the table below:

# Evaluation criteria/Endpoints:

| Instrument | Measurement of interest |
|---|---|
| MoistureMeter D <sup>®</sup> 0.5 mm | Hydration (epidermis + dermis) |
| MoistureMeter D <sup>®</sup> 1.5mm | Hydration (epidermis + dermis) |
| Corneometer® | Hydration (superficial layers of epidermis) |
| Cutometer® | Elasticity |
| Elastimeter® | Elasticity |
| Dermascan® | Skin thickness and density |
| Vivosight OCT® | Skin roughness, density and vascularity |
| Glossymeter® | Brightness |
| Spectrophotometer® | Colour |



| Allergan | Protocol # 18E2581PL | Final version v1.0<br>Date:16/01/2020 |
|---|---|---|
| | Mexameter <sup>®</sup> | Melanin content |
| | Safety Endpoints | |
| | - Injection Site Reactions (ISRs) evaluated by the investigator at each time point after injection. | |
| | - Collection of adverse events and incidents at all visits including severity, action taken, and relationship to device. | |
| | Screening visit: informed consent, medical examination, medical background and previous treatment, subject selection, blood sampling. | |
| Marcha Burana da una sa | | |
| Study Procedures: | | |

| Allergen | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| Allergan | Protocol # 18E2581PL | Date:16/01/2020 |

#### 3. OVERALL STUDY CONSIDERATIONS

#### 3.1. OBJECTIVES

To evaluate the impact on skin quality attributes, including physical measurements following administration of Juvéderm® VOLITE in the volar forearms of healthy volunteers.

#### 3.2. STUDY DESIGN

This study is a prospective, single-center, single arm, open label study in healthy subjects. Each subject will serve as its own control (intra-individual).

#### 3.3. SAMPLE SIZE

This study is an exploratory study, no formal sample size calculation has been performed. 11 subjects will be included to have at least 10 subjects analysed (10% of drop-out rate expected).

#### 3.4. BLINDING

This is an open label study.

#### 3.5. RANDOMIZATION

Not applicable. This is a single-arm study.





| Allorgon | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| Allergan | Protocol # 18E2581PL | Date:16/01/2020 |

#### 3.7. STUDY OUTCOME

#### 3.7.1. Performance outcomes

#### 3.7.1.1. Summary of performance assessments

The table below is a summary of performance parameters.

**Table 2. Summary of performance parameters** 

| Instrument | Measurement of interest | Parameters studied |
|---|---|---|
| MoistureMeter D <sup>®</sup> 0.5 mm | Hydration (epidermis+ dermis) | Hydration rate (TDC) |
| MoistureMeter D <sup>®</sup> 1.5mm | Hydration (epidermis + dermis) | Hydration rate (TDC) |
| Corneometer® | Hydration (superficial layers of epidermis) | Hydration rate (A.U.) |
| Cutometer® | Elasticity | Uf (R0), Ur, Ua (R8), Uf – Ua (R1), Ua/Uf (R2), Ur/Ue (R5), Uv/Ue (R6), Ur/Uf (R7) (mm), Q1, Q2, Q3 |
| Elastimeter® | Elasticity | ISE (N/m) |
| Dermascan <sup>®</sup> | Skin thickness and density | % of non-echogenic surface (skin density), skin thickness (mm) |
| | | For roughness: Ra, Rz |
| Vivosight OCT <sup>®</sup> | Skin roughness, density and vascularity | For density: epidermal thickness, Optical Attenuation Coefficient (OAC) |
| | | For vascularity: plexus depth, vessel diameter, vessel density, density @300 µm |
| Glossymeter® | Brightness | Brightness Index (GU) |
| Spectrophotometer® | Colour | L*, a*, b* (A.U.), ITA°(°) |
| Mexameter® | Melanin content | Melanin Index (A.U.) |

#### 3.7.1.2. Biopsies analysis



Protocol # 18E2581PL Allergan Date:16/01/2020

Final version v1.0



| Allergan | Protocol # 18E2581PL | Final version v1.0<br>Date:16/01/2020 |
|----------|----------------------|---------------------------------------|

#### 3.7.2. Safety outcomes

#### 3.7.2.1. Injection Site Reactions

Immediately after injection, one and three months after injection, the investigator will evaluate the injection site reactions of the tested device with the following 4-point numerical rating scale (NRS):

Table 3. List of ISR

| Parameter | None | Mild | Moderate | Severe |
|-----------------------------|------|------|----------|--------|
| Redness / Erythema | О | | 2 | 3 |
| Pain / Tenderness | О | | 2 | 3 |
| Induration | o | | 2 | 3 |
| Swelling / Oedema | О | | 2 | 3 |
| Lumps / Bumps | О | | 2 | 3 |
| Bruising / Hematoma | О | | 2 | 3 |
| Itching | О | | 2 | 3 |
| Discoloration/ pigmentation | 0 | | 2 | 3 |

Each local reaction will be described by the intensity as follows:

**Table 4. Description of ISR** 

| | Qualification | Definition |
|---|---|---|
| 0 | None | |
| 1 | Mild | Discomfort noted, but no disruption to normal daily activities. No treatment considered |
| 2 | Moderate | Discomfort enough to reduce or affect normal daily activities; treatment may be needed. |
| 3 | Severe | Inability to work or to carry out normal daily activities; treatment is required. |

Moreover, the subjects will be given a daily log in order to grade each ISR described above, each day during 28 days after injection. The ISR will not be reported in the Adverse Event Form excepted if still present at D28, if they require a medical treatment of if judged abnormal by the investigator.

#### 3.7.2.2. Other adverse events

Collection of adverse events by the investigator.



#### 4. STATISTICAL METHODOLOGY

#### 4.1. DESCRIPTIVE ANALYSIS

The quantitative data will be summarized by time point using descriptive statistics:

- Number of values
- Mean
- Median
- Standard deviation (SD)
- Standard error of the mean (SEM)
- First quartile (Q1) and third quartile (Q3)
- Minimum value
- Maximum value

The categorial data will be summarized in frequency (N) and percentage (%).

#### 4.2. LEVEL OF SIGNIFICANCE

All statistical tests will be 2-sided and assessed at  $\alpha = 5\%$  level of significance when applicable.

#### 4.3. STATISTICAL PASS/FAIL CRITERIA TO BE APPLIED

Not applicable, pilot study.

#### 4.4. CRITERIA FOR THE TERMINATION OF THE CLINICAL INVESTIGATION ON STATISTICAL GROUNDS

No statistical criteria have been defined concerning a premature study end.

#### 4.5. DEVIATION(S) FROM THE ORIGINAL STATISTICAL PLAN

Any modification to the statistical analysis plan will be documented as an amendment and will be described in the final study report if applicable.

#### 4.6. ADJUSTMENTS FOR COVARIATES

No covariate is identified for this study, therefore no adjustment for covariates in efficacy analyses is envisaged.

#### 4.7. HANDLING OF DROPOUTS AND MISSING DATA

No strategy for taking in charge missing data has been defined. Data that are not valid or missing will be considered and treated as missing data.

#### 4.8. INTERIM ANALYSES

An analysis will be planned after D94 visit for safety and performance endpoints. A final clinical report will be written after this analysis.

Only a descriptive analysis will be done after the M9 follow-up phone call and a follow-up report will be written.



#### 4.9. MULTIPLE COMPARISONS / MULTIPLICITY

No adjustment for study wise type I error rates will be done.

#### 4.10. EXAMINATION OF SUBGROUPS

No examination of subgroups of patients is planned.

#### 4.11. STATISTICAL SOFTWARE

SAS® 9.4.

#### 5. STATISTICAL ANALYSIS

The study analysis will be performed after the database has been cleaned and judged valid after the blind review meeting. Then, the database will be locked.

#### 5.1. DEFINITION OF ANALYSIS POPULATION

The following analysis populations will be studied and will be considered for the statistical analysis:

- Safety population: any subject having used the tested device.
- FAS (Full Analysis Set): Any subject included in the study with at least a post-basal value.

The analysis of the safety/tolerance parameters will be performed on the "safety" population. The analysis of the performance parameters will be performed on the FAS.

#### 5.2. DESCRIPTIVE STATISTICS

Descriptive statistics will be presented for each parameter. Categorical variables will be summarized with frequency and relative frequency. Continuous variables will be summarized by number of subjects, mean, median, standard deviation, minimum, and maximum. Where appropriate, 2-sided 95% CIs for population mean, or population proportion, will be provided as part of the descriptive summary.

#### **5.3. PATIENT ACCOUNTABILITY**

A flow diagram will be drawn with the number of patients enrolled, the number and % of screen failures and reason for exclusion, the number and % of patients receiving the medical device, the number and % of patients dropping out before and reason for dropping out, and the number and % of patients completing the study.

#### 5.4. DEMOGRAPHIC DATA AND OTHER BASELINE CHARACTERISTICS

The study population will be described on the demographic and injection parameters recorded at the screening and inclusion visits.

The demographic data will be:

- Sex
- Age (variable calculated from birth date and screening visit date)
- Fitzpatrick skin phototype
- Women with childbearing potential
- Contraceptive method



Allergan Protocol # 18E2581PL Final version v1.0
Date:16/01/2020

The injection parameters will be:

- Volume injected
- Injection technique

The listing of medical history and previous and concomitant treatments will also be provided.

#### 5.5. PERFORMANCE EVALUATION

#### 5.5.1. Skin quality measurements

All parameters listed in Table 2 of paragraph 3.7.1.1 ( ) will be analysed using a mixed ANOVA model for repeated measures (MIXED procedure of SAS®) fitted to raw data.

The following factors will be included in the model:

- Zone as fixed (2 levels: treated and control)
- Time as fixed (3 levels: D0, D28 and D84)
- Zone by time interaction
- Subject as random

To capture the correlation between data obtained from a same subject, an unstructured variance -covariance matrix is set.

The following comparisons on adjusted means obtained from the mixed linear model will be performed:

- 1) D28 versus D0 for treated zone
- 2) D84 versus D0 for treated zone
- 3) D84 versus D28 for treated zone
- 4) D28 versus D0 for non-treated zone
- 5) D84 versus D0 for non-treated zone
- 6) D84 vs D28 for non-treated zone
- 7) (D28-D0)treated zone versus (D28-D0)non-treated zone
- 8) (D84-D0)<sub>treated zone</sub> versus (D84-D0)<sub>non-treated zone</sub>
- 9) (D84-D28)treated zone versus (D84-D28)non-treated zone

All adjusted means differences will be tabulated associated with their 95% CI.

The underlying assumptions (residual normality and homoscedasticity) will be analyzed with Shapiro-Wilk test ( $\mathbb{Z}=0.01$ ) and graphs to judge the model validity. In case of strong deviation, a non-parametric approach (Wilcoxon signed rank test) will be carried out.





Allergan

| Allergan | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| | | Date:16/01/2020 |

#### **5.6. SAFETY EVALUATION**

For each parameter of ISR evaluation, the score distribution will be summarized in frequency and percentage by time point.

In addition, for each parameter of ISR evaluation, the proportion of the subjects presenting the sign will be also computed and summarized in frequency and percentage.

At M9, for the safety follow-up phone call, any remarks from the investigator or the subject will be listed.

The individual listing of AE will be provided.

AEs, ADEs, SAEs and SADEs will be summarized by presenting the number and percentage of patients having any sign or symptom. AEs will be classified by System Organ Class (SOCs) and Preferred Term (PTs) using MedDRA.



| Allergan | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| | | Date:16/01/2020 |

## 6. SIGNATURES

SPONSOR: Allergan Pharmaceuticals International Limited



Allergan Protocol # 18E2581PL Final version v1.0
Date:16/01/2020

CRO: Eurofins / Pharmascan



| Allergan | Protocol # 18E2581PL | Final version v1.0 |
|----------|----------------------|--------------------|
| | | Date:16/01/2020 |

# 7. APPENDICES: STRUCTURE OF TABLES

















